CLINICAL TRIAL: NCT01861340
Title: Pilot Study of Lenalidomide and Dexamethasone in Combination With MEDI-551 in Previously Untreated Multiple Myeloma.
Brief Title: Lenalidomide, Dexamethasone and MEDI-551 in Untreated Multiple Myeloma
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: J1340; NA_00081182 (Other: Johns Hopkins)
Record Dates: First submitted 2013-05-20; First posted 2013-05-23 (Estimated); Last update posted 2018-09-10 (Actual); Status verified 2018-09

CONDITIONS: Myeloma
MeSH Terms: conditions — Neoplasms, Plasma Cell | interventions — Lenalidomide; Dexamethasone; inebilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lenalidomide, Dexamethasone, and MEDI-551 (Experimental): Eligible patients will receive Lenalidomide and dexamethasone as per standard of care guidelines for 2 cycles. Patients with a clinical response to lenalidomide and dexamethasone after 2 cycles will proceed to get MEDI-551 for 2 cycles. MEDI-551 will be dosed at 4mg/kg IV on days 1 and 8 of cycle 3 and 4mg/kg IV on day 1 of cycle 4.
  Interventions: Drug: Lenalidomide, Dexamethasone, and MEDI-551

INTERVENTIONS:
Drug: Lenalidomide, Dexamethasone, and MEDI-551 — Patients will receive Lenalidomide and dexamethasone as per standard of care. Patients with a clinical response after 2 cycles will get 2 cycles of MEDI-551.

SUMMARY:
This research study is being done to see if combining the investigational chemotherapy drug, MEDI-551 with the known anti-myeloma drugs, Lenalidomide and Dexamethasone will reduce your myeloma cancer stem cells.

DETAILED DESCRIPTION:
To explore the effect of Lenalidomide, dexamethasone and Medi-551 on multiple myeloma cancer stem cells (CSCs). Myeloma CSCs will be assessed by a clonogenic assay from the bone marrow and flow cytometry from peripheral blood.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 100 years at the time screening
* Symptomatic, previously untreated (with exception of corticosteroids) secretory myeloma
* Written informed consent obtained from the patient/legal representative prior to performing any protocol-related procedures, including screening evaluations
* Patient must agree to take Lenalidomide with low dose dexamethasone as their initial therapy.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
* Life expectancy of >6 months
* Serum creatinine ≤ 2
* ANC≥1000
* Platelets ≥ 50,000
* Total bilirubin ≤ 2 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) ≤ 3 x ULN
* Able to take aspirin (81 or 325 mg) daily as prophylactic anticoagulation (patients intolerant to aspirin may use warfarin or low molecular weight heparin)

Exclusion Criteria:

* Any condition that, in the opinion of the investigator, would interfere with evaluation of the investigational product or interpretation of patient safety or study results.
* Concurrent enrollment in another clinical study, except for non-interventional, observational studies.
* Any chemotherapy, immunotherapy, biologic, investigational, for treatment of multiple myeloma other than Lenalidomide and dexamethasone.
* Previous monoclonal antibody (mAb) or other treatment specifically directed against cluster of differentiation antigen 19 (CD19).
* History of serious allergy or reaction to any component of the MEDI-551 formulation that would prevent administration.
* Previous systemic cancer therapy for myeloma.
* Any active secondary malignancy.
* Human immunodeficiency virus (HIV) positive serology or acquired immune deficiency syndrome.
* Active hepatitis B as defined by seropositivity for hepatitis B surface antigen. Or patients with positive hepatitis B core antibody titers.
* Patients with hepatitis C antibody will be eligible provided that they do not have elevated liver transaminases or other evidence of active hepatitis.
* Documented current central nervous system involvement by multiple myeloma.
* Previous medical history or evidence of an intercurrent illness that may, in the opinion of the investigator, compromise the safety of the patient in the study.
* Diagnosis of plasma cell leukemia
* Diagnosis of POEMS syndrome
* Diagnosis of Amyloidosis
* Diagnosis of non-secretory myeloma

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
The effect of Lenalidomide, dexamethasone and Medi-551 on multiple myeloma cancer stem cells (CSCs). | 16 weeks

SECONDARY OUTCOMES:
The safety of Medi-551 when combined with Lenalidomide and dexamethasone. | 28 weeks

OTHER OUTCOMES:
The pharmacodynamics (reduction in B cells) of this combination | 28 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Carol Ann Huff, MD, Principal Investigator — The Johns Hopkins University
Locations (1):
- The Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No